CLINICAL TRIAL: NCT03919552
Title: Intensity-modulated Radiation Therapy Combined With Cisplatin-based or Carboplatin-based Chemotherapy in Locoregionally Advanced Nasopharyngeal Carcinoma：: A Phase 3 Trial
Brief Title: Cisplatin-based and Carboplatin-based Chemoradiation in Locoregionally Advanced Nasopharyngeal Carcinoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NFEC-2018-013
Record Dates: First submitted 2018-04-25; First posted 2019-04-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Cisplatin; Carboplatin; NPC
Keywords: Nasopharyngeal Carcinoma; cisplatin; carboplatin
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Docetaxel; Carboplatin; Cisplatin

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Carboplatin (Experimental): Patients receive carboplatin (AUC 4 on day 1) every three weeks
  Interventions: Drug: Docetaxel,Carboplatin; Radiation: Carboplatin-based concurrent chemoradiotherapy
- Cisplatin (Active Comparator): Patients receive cisplatin (75mg/m2 on day 1) every three weeks
  Interventions: Drug: Docetaxel,Cisplatin; Radiation: Cisplatin-based concurrent chemoradiotherapy

INTERVENTIONS:
Drug: Docetaxel,Carboplatin — Patients receive docetaxel (75mg/m2 on day 1), carboplatin (AUC 4 on day 1) every three weeks for two cycles before the radiotherapy.
  Other Names: TC induction chemotherapy
  Arms: Carboplatin
Drug: Docetaxel,Cisplatin — Patients receive docetaxel (75mg/m2 on day 1), cisplatin (75mg/m2 on day 1) every three weeks for two cycles before the radiotherapy.
  Other Names: TP induction chemotherapy
  Arms: Cisplatin
Radiation: Carboplatin-based concurrent chemoradiotherapy — Patients receive radical radiotherapy and carboplatin (AUC 5) every three weeks for three cycles during radiotherapy.
  Other Names: Radical radiotherapy and concurrent carboplatin
  Arms: Carboplatin
Radiation: Cisplatin-based concurrent chemoradiotherapy — Patients receive radical radiotherapy and cisplatin (100mg/m2) every three weeks for three cycles during radiotherapy.
  Other Names: Radical radiotherapy and concurrent cisplatin
  Arms: Cisplatin

SUMMARY:
The purpose of this study is to compare cisplatin-based with carboplatin-based chemoradiotherapy in patients with locoregionally advanced nasopharyngeal carcinoma (NPC), in order to confirm the value of carboplatin-based chemoradiotherapy in NPC patients.

DETAILED DESCRIPTION:
Patients presented with non-keratinizing NPC and stage T3-4NxM0/TxN2-3M0 are randomly assigned to receive cisplatin-based (control arm) with carboplatin-based (investigational arm) chemoradiotherapy. Patients in the investigational arm receive docetaxel (75mg/m2 on day 1), carboplatin (AUC 4 on day 1) every three weeks for two cycles before the radiotherapy, and then receive radical radiotherapy and carboplatin (AUC 5 on day 1) every three weeks for three cycles during radiotherapy. Patients in the control arm receive docetaxel (75mg/m2 on day 1), cisplatin (75mg/m2 on day 1) every three weeks for two cycles before the radiotherapy, and then receive radical radiotherapy and cisplatin (100mg/m2 on day 1) every three weeks for three cycles during radiotherapy. Patients are stratified according to stage. The primary end point is overall survival (OS). Secondary end points include failure-free survival (FFS), distant failure-free survival (D-FFS), locoregional failure-free survival (LR-FFS), initial response rates after treatments and toxic effects. All efficacy analyses are conducted in the intention-to-treat population; the safety population include only patients who receive their randomly assigned treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly histologically confirmed non-keratinizing (according to World Health Organization (WHO) histologically type).
* Tumor staged as T3-4Nx/TxN2-3 (according to the 8th American Joint Commission on Cancer edition).
* No evidence of distant metastasis (M0).
* Satisfactory performance status: Karnofsky scale (KPS) > 70.
* Adequate marrow: leucocyte count ≥4000/μL, hemoglobin ≥90g/L and platelet count ≥100000/μL.
* Normal liver function test: Alanine Aminotransferase (ALT)、Aspartate Aminotransferase (AST) <1.5×upper limit of normal (ULN) concomitant with alkaline phosphatase (ALP) ≤2.5×ULN, and bilirubin ≤ULN.
* Adequate renal function: creatinine clearance ≥60 ml/min.
* Patients must be informed of the investigational nature of this study and give written informed consent.

Exclusion Criteria:

* WHO Type keratinizing squamous cell carcinoma or basaloid squamous cell carcinoma.
* Age ≥65 years or <18 years.
* Treatment with palliative intent.
* Prior malignancy except adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer.
* Pregnancy or lactation.
* History of previous radiotherapy (except for non-melanomatous skin cancers outside intended RT treatment volume).
* Prior chemotherapy or surgery (except diagnostic) to primary tumor or nodes.
* Any severe intercurrent disease, which may bring unacceptable risk or affect the compliance of the trial, for example, unstable cardiac disease requiring treatment, renal disease, chronic hepatitis, diabetes with poor control (fasting plasma glucose >1.5×ULN), and emotional disturbance.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 482 (Estimated)
Dates: Start 2018-01-31 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Failure-free survival | 3-year
  Failure-free survival is calculated from the date of randomisation to the date of treatment failure or death from any cause, whichever is first.

SECONDARY OUTCOMES:
Locoregional failure-free survival | 3-year
  Locoregional failure-free survival is calculated from randomisation to the first locoregional failure.
Distant failure-free survival | 3-year
  Distant failure-free survival is calculated from randomisation to the first locoregional failure.
The initial response rates after treatments | A week after completion of the last cycle of induction chemotherapy and 16 weeks after completion of radiotherapy.
  The initial response rates is calculated at the time 1 week after completion of the last cycle of induction chemotherapy and 16 weeks after completion of radiotherapy.
Toxic effects | 3-year
  Radiation and chemotherapy related toxic effects as assessed by CTCAE v4.0.
Overall survival | 3-year
  Overall survival is calculated from randomization to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Jian Guan, Study Chair — Nanfang Hospital, Southern Medical University
Locations (1):
- Southern medical university, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Haddad RI, Shin DM. Recent advances in head and neck cancer. N Engl J Med. 2008 Sep 11;359(11):1143-54. doi: 10.1056/NEJMra0707975. No abstract available. PMID 18784104
- [Background] Guan J, Zhang Y, Li Q, Zhang Y, Li L, Chen M, Xiao N, Chen L. A meta-analysis of weekly cisplatin versus three weekly cisplatin chemotherapy plus concurrent radiotherapy (CRT) for advanced head and neck cancer (HNC). Oncotarget. 2016 Oct 25;7(43):70185-70193. doi: 10.18632/oncotarget.11824. PMID 27602493
- [Background] Hashibe M, Brennan P, Chuang SC, Boccia S, Castellsague X, Chen C, Curado MP, Dal Maso L, Daudt AW, Fabianova E, Fernandez L, Wunsch-Filho V, Franceschi S, Hayes RB, Herrero R, Kelsey K, Koifman S, La Vecchia C, Lazarus P, Levi F, Lence JJ, Mates D, Matos E, Menezes A, McClean MD, Muscat J, Eluf-Neto J, Olshan AF, Purdue M, Rudnai P, Schwartz SM, Smith E, Sturgis EM, Szeszenia-Dabrowska N, Talamini R, Wei Q, Winn DM, Shangina O, Pilarska A, Zhang ZF, Ferro G, Berthiller J, Boffetta P. Interaction between tobacco and alcohol use and the risk of head and neck cancer: pooled analysis in the International Head and Neck Cancer Epidemiology Consortium. Cancer Epidemiol Biomarkers Prev. 2009 Feb;18(2):541-50. doi: 10.1158/1055-9965.EPI-08-0347. Epub 2009 Feb 3. PMID 19190158
- [Background] Blot WJ, McLaughlin JK, Winn DM, Austin DF, Greenberg RS, Preston-Martin S, Bernstein L, Schoenberg JB, Stemhagen A, Fraumeni JF Jr. Smoking and drinking in relation to oral and pharyngeal cancer. Cancer Res. 1988 Jun 1;48(11):3282-7. PMID 3365707
- [Background] Chang ET, Adami HO. The enigmatic epidemiology of nasopharyngeal carcinoma. Cancer Epidemiol Biomarkers Prev. 2006 Oct;15(10):1765-77. doi: 10.1158/1055-9965.EPI-06-0353. PMID 17035381
- [Background] Klein G. Nasopharyngeal carcinoma (NPC) is an enigmatic tumor. Semin Cancer Biol. 2002 Dec;12(6):415-8. doi: 10.1016/s1044579x02000834. No abstract available. PMID 12450726
- [Background] Buell P. The effect of migration on the risk of nasopharyngeal cancer among Chinese. Cancer Res. 1974 May;34(5):1189-91. No abstract available. PMID 4842361
- [Background] Ozer E, Grecula JC, Agrawal A, Rhoades CA, Young DC, Schuller DE. Long-term results of a multimodal intensification regimen for previously untreated advanced resectable squamous cell cancer of the oral cavity, oropharynx, or hypopharynx. Laryngoscope. 2006 Apr;116(4):607-12. doi: 10.1097/01.mlg.0000208340.42071.f9. PMID 16585867
- [Background] Fallai C, Bolner A, Signor M, Gava A, Franchin G, Ponticelli P, Taino R, Rossi F, Ardizzoia A, Oggionni M, Crispino S, Olmi P. Long-term results of conventional radiotherapy versus accelerated hyperfractionated radiotherapy versus concomitant radiotherapy and chemotherapy in locoregionally advanced carcinoma of the oropharynx. Tumori. 2006 Jan-Feb;92(1):41-54. doi: 10.1177/030089160609200108. PMID 16683383
- [Background] Blanchard P, Baujat B, Holostenco V, Bourredjem A, Baey C, Bourhis J, Pignon JP; MACH-CH Collaborative group. Meta-analysis of chemotherapy in head and neck cancer (MACH-NC): a comprehensive analysis by tumour site. Radiother Oncol. 2011 Jul;100(1):33-40. doi: 10.1016/j.radonc.2011.05.036. Epub 2011 Jun 16. PMID 21684027
- [Background] Sun Y, Li WF, Chen NY, Zhang N, Hu GQ, Xie FY, Sun Y, Chen XZ, Li JG, Zhu XD, Hu CS, Xu XY, Chen YY, Hu WH, Guo L, Mo HY, Chen L, Mao YP, Sun R, Ai P, Liang SB, Long GX, Zheng BM, Feng XL, Gong XC, Li L, Shen CY, Xu JY, Guo Y, Chen YM, Zhang F, Lin L, Tang LL, Liu MZ, Ma J. Induction chemotherapy plus concurrent chemoradiotherapy versus concurrent chemoradiotherapy alone in locoregionally advanced nasopharyngeal carcinoma: a phase 3, multicentre, randomised controlled trial. Lancet Oncol. 2016 Nov;17(11):1509-1520. doi: 10.1016/S1470-2045(16)30410-7. Epub 2016 Sep 27. PMID 27686945
- [Background] Blanchard P, Lee A, Marguet S, Leclercq J, Ng WT, Ma J, Chan AT, Huang PY, Benhamou E, Zhu G, Chua DT, Chen Y, Mai HQ, Kwong DL, Cheah SL, Moon J, Tung Y, Chi KH, Fountzilas G, Zhang L, Hui EP, Lu TX, Bourhis J, Pignon JP; MAC-NPC Collaborative Group. Chemotherapy and radiotherapy in nasopharyngeal carcinoma: an update of the MAC-NPC meta-analysis. Lancet Oncol. 2015 Jun;16(6):645-55. doi: 10.1016/S1470-2045(15)70126-9. Epub 2015 May 6. PMID 25957714
- [Background] Munro AJ. An overview of randomised controlled trials of adjuvant chemotherapy in head and neck cancer. Br J Cancer. 1995 Jan;71(1):83-91. doi: 10.1038/bjc.1995.17. PMID 7819055
- [Background] Akhlaghi F, Esmaeelinejad M, Shams A, Augend A. Evaluation of neo-adjuvant, concurrent and adjuvant chemotherapy in the treatment of head and neck squamous cell carcinoma: a meta-analysis. J Dent (Tehran). 2014 May;11(3):290-301. Epub 2014 May 31. PMID 25628664